CLINICAL TRIAL: NCT05785039
Title: Phase IIa/IIb Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of BL-B01D1 for Injection in Patients With Multiple Solid Tumors, Including Locally Advanced or Metastatic Urinary System Tumors
Brief Title: A Study of BL-B01D1 in Patients With Multiple Solid Tumors, Including Locally Advanced or Metastatic Urinary System Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-201
Record Dates: First submitted 2023-03-09; First posted 2023-03-27 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Urinary System Tumor; Solid Tumor
MeSH Terms: conditions — Urologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive BL-B01D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507

SUMMARY:
Phase IIa/IIb clinical study to evaluate the safety, tolerability, pharmacokinetics and efficacy of BL-B01D1 for injection in patients with multiple solid tumors such as locally advanced or metastatic urinary system tumors.

DETAILED DESCRIPTION:
Phase IIa: To explore the safety and initial efficacy of BL-B01D1 in a variety of solid tumors such as locally advanced or metastatic urinary system tumors, and further determine RP2D. The preliminary efficacy, pharmacokinetic characteristics and immunogenicity of BL-B01D1 were evaluated. Phase IIb: To explore the efficacy of BL-B01D1 as a single agent RP2D obtained in a Phase IIa clinical study. To evaluate the safety and tolerability, pharmacokinetic characteristics and immunogenicity of BL-B01D1.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily and follow the protocol requirements;
2. Gender is not limited;
3. Age: ≥18 years old and ≤75 years old;
4. Expected survival time ≥3 months;
5. Locally advanced or metastatic urothelial carcinoma and other solid tumors confirmed by histopathology and/or cytology after failure or intolerance to standard treatment or for which standard treatment is currently unavailable or unavailable;
6. Testosterone levels in prostate cancer < 1.73 nmol/L (50 ng/dL), disease progression before screening, according to the PCWG3 consensus;
7. Agree to provide archived tumor tissue samples or fresh tissue samples of primary or metastatic lesions within 3 years. If the subjects cannot provide tumor tissue samples, they can be enrolled after the evaluation of the investigators if they meet other inclusion and exclusion criteria;
8. At least one measurable lesion (other than prostate cancer), as defined by RECIST v1.1, was required;
9. ECOG 0 or 1;
10. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 defined by NCI-CTCAE v5.0;
11. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
12. With adequate organ function;
13. For premenopausal women who are likely to have children, a pregnancy test must be performed within 7 days before starting treatment, a serum or urine pregnancy test must be negative, and the patient must not be lactating; All enrolled patients (male or female) were advised to use adequate barrier contraception throughout the treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Antineoplastic therapy within 4 weeks or 5 half-lives before the first dose; Mitomycin and nitrosoureas were administered within 6 weeks before the first dose; Oral fluorouracil drugs;
2. History of severe cardiovascular and cerebrovascular diseases;
3. Prolonged QT interval, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
4. Active autoimmune and inflammatory diseases;
5. Other malignant tumors that progressed or required treatment within 5 years before the first dose;
6. Patients with poor blood glucose control before the first dose;
7. Hypertension poorly controlled with two antihypertensive drugs before the first dose or previous history of hypertensive crisis or hypertensive encephalopathy;
8. A history of interstitial lung disease (ILD), current ILD, or suspicion of such disease on imaging during screening;
9. Complicated with pulmonary diseases leading to clinically severe respiratory function impairment;
10. Were receiving &gt before the first dose; Long-term systemic corticosteroid therapy with 10mg/ day prednisone or equivalent anti-inflammatory active drugs or any form of immunosuppressive therapy;
11. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening;
12. Patients with central nervous system (CNS) metastases and/or carcinomatous meningitis (meningeal metastases) and/or spinal cord compression;
13. Patients with massive or symptomatic effusions or poorly controlled effusions;
14. Imaging examination indicated that the tumor had invaded or wrapped the large blood vessels of the chest, neck, and pharynx, except that the investigator thought that it would not affect the patient's enrollment in the drug;
15. Patients with a history of allergy to recombinant humanized antibody or human-mouse chimeric antibody or to any of BL-B01D1's excipients;
16. Prior organ transplantation or allogeneic hematopoietic stem cell transplantation;
17. Human immunodeficiency virus antibody positive, active tuberculosis, active hepatitis B virus infection or active hepatitis C virus infection;
18. Had a serious infection within 4 weeks before the first dose of study drug; Indications of active pulmonary infection within 2 weeks before the first dose of study drug;
19. Patients with superior vena cava syndrome should not be rehydrated;
20. Had a history of severe neurological or psychiatric disorders;
21. Imaging examination showed that the tumor had invaded or wrapped the large thoracic vessels;
22. Serious unhealed wounds, ulcers, or fractures, or clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
23. Subjects scheduled to receive live vaccine or within 28 days before the first dose;
24. Other circumstances that the investigator deemed inappropriate for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase IIa: Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-B01D1.
Phase IIb: Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.

SECONDARY OUTCOMES:
Phase IIa/IIb: Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.
Phase IIa: Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Phase IIb: Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of BL-B01D1 to the first date of either disease progression or death, whichever occurs first.
Phase IIa/IIb: Disease control rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Phase IIa/IIb: Duration of response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Phase IIa/IIb: Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of BL-B01D1 will be investigated.
Phase IIa/IIb: Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of BL-B01D1 will be investigated.
Phase IIa: T1/2 | Up to approximately 24 months
  Half-life (T1/2) of BL-B01D1 will be investigated.
Phase IIa: AUC0-t | Up to approximately 24 months
  Blood concentration - Area under time line.
Phase IIa: CL | Up to approximately 24 months
  To study the serum clearance rate of BL-B01D1 per unit time.
Phase IIa/IIb: Ctrough | Up to approximately 24 months
  Ctrough is defined as the lowest serum concentration of BL-B01D1 prior to the next dose will be administered.
Phase IIa/IIb: Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency and titer of anti-BL-B01D1 antibody (ADA) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, PHD, Principal Investigator — Fudan University
Locations (1):
- Fudan University ShangHai Cancer Center, Shanghai, Shanghai Municipality, China